CLINICAL TRIAL: NCT07406178
Title: JY509 Universal NK Cell Injection for the Treatment of Relapsed or Refractory Pediatric B-cell Acute Lymphoblastic Leukemia
Brief Title: JY509 Universal NK Cell Injection for the Treatment of Relapsed/Refractory Pediatric B-ALL
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025137
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Relapsed/Refractory Pediatric B-ALL
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JY509 universal NK cell injection (Experimental)
  Interventions: Biological: JY509 universal NK cell injection

INTERVENTIONS:
Biological: JY509 universal NK cell injection — 3+3 dose escalation trial and dose expansion trial

SUMMARY:
This is a single-arm, open-label, dose-escalation and expansion, prospective clinical trial conducted in patients with relapsed or refractory pediatric B-cell acute lymphoblastic leukemia to evaluate the safety and efficacy of JY509 universal NK cell injection.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as relapsed or refractory B-cell acute lymphoblastic leukemia (B-ALL), and meeting any of the following criteria:①The patient fails to achieve bone marrow complete remission (MRD > 1%) after at least 2 courses of standard induction chemotherapy; or those with pre-treatment specific molecular markers/immunophenotypes do not achieve molecular/immunological complete remission (remain non-negative post-treatment);②Relapse during chemotherapy, early relapse within 12 months after treatment discontinuation, or late relapse ≥ 12 months after complete remission, with failure to achieve complete remission (MRD > 1%) following 1 course of standard induction chemotherapy;③Relapsed after hematopoietic stem cell transplantation (HSCT);④Isolated bone marrow relapse, isolated extramedullary relapse (testicular leukemia, central nervous system leukemia), or combined relapse;
* Tumor cells confirmed positive for CD19 by flow cytometry (FCM) or immunohistochemistry (IHC);
* Expected survival ≥ 3 months from the date of signing the informed consent form (ICF);
* Aged 3-18 years (inclusive), no gender restriction;
* ECOG ≤ 2;
* HGB ≥ 70 g/L, PLT ≥ 50×10⁹/L (recombinant human erythropoietin or blood transfusion permitted);
* Liver and kidney functions, as well as cardiopulmonary functions, shall meet the following requirements:①LVEF≥50%;②Oxygen saturation ≥ 90%;③Total bilirubin ≤3×ULN;④ALT/AST<3×ULN;⑤Serum creatinine≤2×ULN.If organ dysfunction links to the disease, investigator evaluates enrollment;
* The subject or guardian understands and signs the informed consent form.

Exclusion Criteria:

* Severe cardiac or pulmonary insufficiency, which the investigator deems inappropriate for enrollment.
* Complicated with other progressive malignant tumors.
* Presence of active and/or uncontrolled infections that have not been effectively managed.
* Complicated with severe autoimmune diseases or congenital immunodeficiency.
* Subjects to be excluded if: testing positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) at screening, with peripheral blood hepatitis B virus (HBV) DNA levels above the lower limit of detection; testing positive for hepatitis C virus (HCV) antibody, with positive peripheral blood HCV RNA; testing positive for human immunodeficiency virus (HIV) antibody; testing positive for Treponema pallidum particle agglutination assay (TPPA).
* A history of severe hypersensitivity to biological products (including antibiotics).
* Patients who have undergone allogeneic hematopoietic stem cell transplantation and still suffer from acute graft-versus-host disease (GVHD) one month after discontinuation of immunosuppressive agents.
* Unstable systemic diseases as judged by the investigator, including but not limited to severe hepatic, renal or metabolic diseases requiring drug therapy.
* Having received major surgery assessed by the investigator as unsuitable for enrollment within 4 weeks prior to screening.
* Patients with other severe physical or mental diseases or abnormal laboratory test results that may increase the risk of study participation or interfere with study outcomes, as well as those who are deemed unsuitable for participation in this study by the investigator.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence frequency, number of cases,incidence rate and severity of adverse events and adverse reactions occurring after infusion and before withdrawal or the safety follow-up period. | From enrolment to one year after infusion